CLINICAL TRIAL: NCT06801639
Title: Advancing Alzheimer's Care: Home-based tDCS (Transcranial Direct Current Stimulator) for Affective Symptoms
Brief Title: Advancing Alzheimer's Care: Home-based tDCS for Affective Symptoms
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center at San Antonio (Other)
Collaborators: Alzheimer's Association (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: STUDY00001032
Record Dates: First submitted 2025-01-24; First posted 2025-01-30 (Actual); Last update posted 2026-02-11 (Actual); Status verified 2026-02

CONDITIONS: Alzheimer Disease
Keywords: Transcranial direct current stimulation; TDCS; Home-based; Cognitive symptoms
MeSH Terms: conditions — Alzheimer Disease; Neurobehavioral Manifestations | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: This is a randomized double-blind cross-over clinical trial to investigate the effects of transcranial direct current stimulation (tDCS) over affective symptoms (AS) of patients with Alzheimer's disease (AD). The study will also investigate underlying neurobiological mechanisms of tDCS in AD with functional and structural neuroimaging techniques.
Who Masked: Participant, Investigator
Masking Description: Patients will be blinded throughout the trial. As the application of tDCS electrical current over the skin can be perceived by the participants, the study team will employ a sham condition that has been shown to be reliable and indistinguishable from active treatment in previous clinical trials published in the available scientific literature. An individual on the study team will be delegated to randomize and program and re-program devices. Participants will act as their own control. The researcher supervising the stimulation will be blinded to the intervention the participant is receiving.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Active TDCS treatment (Experimental): The active-tDCS treatment will consist of a constant 2mA current applied during 30-minute sessions with a 30 second ramp up and ramp down at the start and end of the stimulation.
  Interventions: Device: Transcranial direct current stimulation (tDCS)
- Sham TDCS treatment (Sham Comparator): Sham-tDCS treatment will consist of the same montage as the active TDCS with the built-in function of the device that has been shown to be indistinguishable from the active treatment in previous trials described in the literature.
  Interventions: Device: Sham tDCS

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) — The active-tDCS treatment will consist of a constant 2mA current applied during daily 30-minute sessions with a 30 second ramp up and ramp down at the start and end of the stimulation. The anode electrode will be placed over the left dorsolateral prefrontal cortex (DLPFC) and the cathode electrode over the right DLPFC.
  Other Names: tDCS
  Arms: Active TDCS treatment
Device: Sham tDCS — Sham-tDCS treatment will consist of the same montage as the active TDCS with the built-in function of the device that has been shown to be indistinguishable from the active treatment in previous trials described in the literature.
  Other Names: Control
  Arms: Sham TDCS treatment

SUMMARY:
Participants will be asked to participate in this research study of a device that creates transcranial direct current stimulation (tDCS).

The researchers hope to learn if 30 minute sessions of transcranial direct current stimulation (tDCS) improve such a mood or feelings in people with Alzheimer's Disease.

This study involves the use of an investigational device called a tDC stimulator. "Investigational" means that the device has not yet been approved by the U.S. Food & Drug Administration (FDA) for treating Alzheimer's Disease.

This study will help find out what effects, good and/or bad, this has. The safety of this device in humans has been tested in prior research studies; however, some side effects may not yet be known.

DETAILED DESCRIPTION:
Three in-person visits will occur: (1) on the week prior to the first day of stimulation visit patients will undergo brain MRI scan to collect T1, T2, DWI and resting state functional MRI (rs-fMRI), and functional Near-Infrared Spectroscopy/Electroencephalography (fNIRS/EEG) imaging. In this visit, patients and caregivers will be taught how to operate the tDCS device and will receive a unit to take home; (2) on the day after completing the first treatment period, patients will undergo a second MRI scan with the same sequences and fNIRS/EEG imaging; (3) on the day after completing the second treatment period, at the end of week 5, patients will return the tDCS device to the study team and perform a last fNIRS/EEG imaging.

At in-person visits and during treatment periods patients will be asked questions regarding tolerability and acceptability, including monitoring for side effects, as well as completing questionnaires that assess cognition and NPS. All sessions will be remotely supervised via video conference platform.

ELIGIBILITY:
Inclusion Criteria:

1. Ability of subject to understand and the willingness to sign a written informed consent document.
2. Individuals who are 60 years or older.
3. Diagnosis of possible or probable AD according to the National Institute of Aging - Alzheimer's Association diagnostic criteria; individuals with mild cognitive impairment (MCI) due to AD, as defined by these criteria, are eligible if biomarker evidence supports the underlying AD pathology (e.g., amyloid or tau positivity in CSF or PET imaging).
4. In the determination of the PI in consultation with the delegated physician(s) patient's signs/symptoms are consistent with: a Clinical Dementia Rating (CDR) of 0.5 (MCI) with biomarker evidence of AD; or a Clinical Dementia Rating score of 1-2 (mild to moderate dementia).
5. Clinically meaningful AS of ADRD is defined by the presence of any affective symptom (i.e., depression, elation, anxiety, irritability, and apathy) and a total severity score on the NPI-Q ≥10.
6. Have an eligible caregiver willing to be present during stimulation sessions and answer questionnaires (see criteria below).
7. Can speak and read in English.
8. Stable doses of medications for at least one month.
9. Access to a reliable broadband internet connection.

Caregiver

1. An adult who serves as an unpaid caregiver for an individual enrolled in the study as interpreted by the PI or delegate physician.
2. Adequate cognitive capacity to provide verbal consent to participate in the caregiver arm of the study.
3. Adequate reading, writing, hearing and verbal capacity to provide collateral information about the study participant, answer questions related to their health and care, and assist in tDCS sessions,

Exclusion Criteria:

1. Unstable medical conditions (e.g. unstable angina, uncontrolled diabetes and hypertension, advanced cancer, etc.) that, in the opinion of the PI in consultation with delegated physician(s) would contraindicate study participation for safety or data quality reasons.
2. Medical history of serious psychiatric disorders (i.e. bipolar disorder, schizophrenia, manic depression etc.).
3. History of epilepsy.
4. Metallic objects in the brain, skull, or otherwise placed where it could interfere with DCS.
5. Have risk of suicidal behavior, defined as any suicidal behavior or suicidal ideation of type 4 (active suicidal ideation with some intent to act, without specific plan) or type 5 (active suicidal ideation with specific plan and intent) based on the Columbia-Suicide Severity Rating Scale (C-SSRS) in the 3 months prior to screening;
6. Unwillingness to undergo MRI at baseline and during the Week 2 conversion period for reasons other than a confirmed medical contraindication such as having a pacemaker or other implanted medal making MRI unsafe.
7. Being an active participant in other therapeutic clinical trial.

Caregiver

1. Any individual who does not meet all the inclusion criteria

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2025-07-15 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2028-12 (Estimated)

PRIMARY OUTCOMES:
Neuropsychiatric Inventory Questionnaire (NPI-Q) severity score | Baseline to Day 35
  A 12 item questionnaire that measures a broad range of psychiatric symptoms. Each individual item is scored from 0 to 3.
  Total scores range from 0 to 36, with higher scores indicating more severe symptoms.
Brief Dimensional Apathy Scale (bDAS) | Baseline to Day 35
  A 9 item scale completed by caregivers about the participant. Each item is scored from 0 to 3.
  Total scores range from 0-27 with a higher score indicating more severe apathy.
Caregiver version of the Irritability Questionnaire (IrQ) How often | Baseline to Day 35
  A 10 item questionnaire, and each item is scored from 0 to 3. Total scores can range from 0-30 with a higher score indicating more frequent symptoms.
Caregiver version of the Irritability Questionnaire (IrQ) How much | Baseline to Day 35
  A 10 item questionnaire, and each item is scored from 0 to 3. Total scores can range from 0-30 with a higher score indicating more severe symptoms.
Cornell Scale for Depression in Dementia (CSDD) | Baseline to Day 35
  A 19 item scale which is scored as follows:
  a - Unable to evaluate the sign or symptom 0 - Absent
  1. - Mild or intermittent
  2. - Severe Total scores range from 0-38 with a higher score indicating greater depression.
Generalized Anxiety Disorder-7 Scale (GAD-7) | Baseline to Day 35
  A 7 item scale scored as follows:
  0 - Not at all
  1. - Several days
  2. - More than half the days
  3. - Nearly every day Total scores range from 0-21 with a higher score indicating greater anxiety.
Montreal Cognitive Assessment (MoCA) | Baseline to Day 35
  A battery of cognitive assessment tasks. Total possible score that can be achieved is between 0-30. A higher score indicating better cognition.

CONTACTS AND LOCATIONS:
Overall Officials: Thiago Macedo e Cordeiro, MD, MSc, Principal Investigator — The University of Texas Health Science Center at San Antonio
Locations (1):
- University of Texas Health Science Center at San Antonio, San Antonio, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
Data collected for this study will be analyzed and stored at the Glenn Bigs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio. After the study is completed, the de-identified, archived data will be transmitted to and stored at the Glenn Bigs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio, for use by other researchers including those outside of the study. Permission to transmit data to the Glenn Biggs Institute for Alzheimer's and Neurodegenerative diseases at UT Health San Antonio will be included in the informed consent.
Supporting Information: Study Protocol, SAP
Time Frame: When the study is completed and data is analyzed.